CLINICAL TRIAL: NCT05755178
Title: Music, Feelings and Relationships - Implementation and Evaluation of a Group Intervention for Children in Shelters
Brief Title: Musical Group Intervention for Children in Shelters
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Kronoberg County Council (Other Government)
Collaborators: Musik i Syd (Unknown); Kvinnojouren Blenda (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MGSB
Record Dates: First submitted 2023-02-12; First posted 2023-03-06 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-10

CONDITIONS: Domestic Violence; Child Development; Psychological Distress; Music Therapy; Group Intervention

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Musical group intervention (Experimental): A music group intervention, offered to children 3-10 years who live or have lived at a shelter.
  6 group sessions with musicians and music therapist and a group of 4-8 children.
  Focus on improving recognition and regulation of emotions, and on relational capacity with adults and peers.
  Interventions: Behavioral: Music, feelings and relationships - music group for children at shelters

INTERVENTIONS:
Behavioral: Music, feelings and relationships - music group for children at shelters — A music group intervention, offered to children 3-10 years who live or have lived at a shelter.
  6 group sessions with musicians and music therapist and a group of 4-8 children.
  Focus on improving recognition and regulation of emotions, and on relational capacity with adults and peers.

SUMMARY:
The aim of the study is to augment knowledge on interventions for children who live, or have lived, in shelters after exposure to domestic violence. Research questions concern the feasibility of a music group intervention for children. The experiences of children, caregivers, and professionals will be investigated. Additionally, outcomes concerning emotional reactivity, capacity for emotional regulation, quality of life, and psychological health will be evaluated.

DETAILED DESCRIPTION:
Research problem and specific questions The project uses a mixed methods design in a naturalistic setting. Qualitative data concerning how children, caregivers and professionals experience the intervention and quantitative data concerning practical feasibility, adaptions made, and children's reported psychological health and quality of life will be studied. Data will be collected through questionnaires, log-forms, evaluation forms, and interviews with children, parents, and professionals. Thematic analysis and Interpretative phenomenological analysis will be used for qualitative data. Descriptive statistics and non-parametric methods will be used as applicable for quantitative data.

Plan for project realization The music group intervention will be offered to children 3-10 years, who live or have lived at a shelter. In all 12 groups with 4-8 children in each (48-96 children) will be realized. Collaboration with 2-3 shelters is established.

Questionnaires designed to measure psychological health, health-related quality of life, emotion reactivity, and capacity for emotional regulation will be administrated to caregivers pre- and post-intervention. A log-form will be filled out by professionals after each group session. Evaluation forms will be administrated to children, caregivers, and professionals after completing the intervention. Qualitative interviews focusing on feasibility, acceptance, and experiences of the intervention will be carried through with children, caregivers and professionals post intervention.

ELIGIBILITY:
Inclusion Criteria:

* Age 3-10 years
* Currently living or have lived at shelter together with a caregiver

Ages: 3 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 96 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline on Strengths and Difficulties Questionnaire - Parent version at termination of intervention. | Up to 4 months
  Caregiver report of child psychopathology. Minimum score 0, maximum score 40, higher score indicating worse outcome.
Change from baseline on Child Healthy Utility 9D at termination of intervention. | Up to 4 months
  Caregiver report of child health related quality of life. Minimum score 0, maximum score 36, higher score indicating worse outcome.
Change from baseline on Emotion Questionnaire for parents at termination of intervention. | Up to 4 months
  Caregiver report of child health related quality of life. Minimum score 0, maximum score 36135, higher score indicating worse outcome.

SECONDARY OUTCOMES:
Evaluation form Music group for children at shelters - child version | Up to 4 months
  Scores and free text answers on satisfaction and experiences of participating in the intervention.
Evaluation form Music group for children at shelters - parent version | Up to 4 months
  Scores and free text answers on parental satisfaction and experiences after havein a child participating in the intervention.
Evaluation form Music group for children at shelters - professional version | Up to 4 months
  Scores and free text answers on satisfaction and experiences of participating in the intervention.

OTHER OUTCOMES:
Feasibility of the intervention Music group for children at shelters. | Up to 4 months
  Log after each session on participation and adaptions made.
Childrens' experiences of participating in Music group for children at shelters. | Up to 4 months
  Qualitative data from interviews with children.
Parents' experiences of having a child participating in Music group for children at shelters. | Up to 4 months
  Qualitative data from interviews with parents.
Professionals' experiences of participating in Music group for children at shelters. | through study completion, an average of 2 years
  Qualitative data from interviews with professionals taking part in the intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Research and Development, Region Kronoberg, Vaxjo, Sweden

IPD SHARING:
Plan to Share IPD: No